CLINICAL TRIAL: NCT04815551
Title: A Phase 1, First-in-human, Randomized, Placebo Controlled, Double Blind, Single Ascending Dose (SAD) Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Immunogenicity of AV-380 in Healthy Subjects
Brief Title: A Phase 1 Study of AV-380 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AV-380-20-101
Record Dates: First submitted 2021-03-08; First posted 2021-03-25 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Cachexia
MeSH Terms: conditions — Cachexia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- AV-380 IV 4 mg/kg (Experimental): IV infusion of AV-380 at dose level 4 mg/kg
  Interventions: Drug: AV-380
- AV-380 IV 8 mg/kg (Experimental): IV infusion of AV-380 at dose level 8 mg/kg
  Interventions: Drug: AV-380
- AV-380 IV 13 mg/kg (Experimental): IV infusion of AV-380 at dose level 13 mg/kg
  Interventions: Drug: AV-380
- AV-380 IV 20 mg/kg (Experimental): IV infusion of AV-380 at dose level 20 mg/kg
  Interventions: Drug: AV-380
- AV-380 SC 4 mg/kg (Experimental): Subcutaneous injection of AV-380 at dose level 4 mg/kg
  Interventions: Drug: AV-380
- AV-380 SC 2 mg/kg (Experimental): Subcutaneous injection of AV-380 at dose level 2 mg/kg
  Interventions: Drug: AV-380
- AV-380 SC 1 mg/kg (Experimental): Subcutaneous injection of AV-380 at dose level 1 mg/kg
  Interventions: Drug: AV-380
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AV-380 — AV-380 is an immunoglobulin (Ig) G1 monoclonal antibody (mAb) intended to bind circulating human growth differentiation factor 15 (GDF-15), a cytokine involved in cancer-induced cachexia.
  Arms: AV-380 IV 13 mg/kg; AV-380 IV 20 mg/kg; AV-380 IV 4 mg/kg; AV-380 IV 8 mg/kg; AV-380 SC 1 mg/kg; AV-380 SC 2 mg/kg; AV-380 SC 4 mg/kg
Drug: Placebo — Placebo is sterile liquid for IV infusion.
  Arms: Placebo

SUMMARY:
This double-blinded, placebo-controlled, single ascending dose (SAD) study is designed to evaluate the safety, pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity in healthy subjects of a single dose of AV-380. AV-380 is an immunoglobulin (Ig) G1 monoclonal antibody (mAb) intended to bind circulating human growth differentiation factor 15 (GDF-15), a cytokine involved in cancer-induced cachexia.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female volunteers, 18 to 50 years of age, inclusive.
2. A body mass index (BMI) between 18 and 30 kg/m2 and weight between 60 and 90 kg.
3. Healthy as indicated by a comprehensive clinical assessment (detailed medical history and complete physical examination). Supine blood pressure (BP), heart rate (HR), electrocardiogram (ECG) intervals and routine laboratory tests within the normal range of the study center (see Appendix 4) or considered not clinically significant by the Investigator. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and total bilirubin must be < 1.5 times the upper limit of the normal range (ULN). Total bilirubin, if above 1.5 x ULN, is only acceptable with a history of Gilbert's Syndrome.
4. Non-smoker or ex-smoker for longer than 6 months.
5. Sexually active pre-menopausal female subjects and female partners of male subjects must use adequate contraceptive measures, while on study and for at least 100 days after the IMP administration. Sexually active male subjects must use adequate contraceptive measures, while on study and for at least 160 days after the last dose of IMP. All fertile male and female subjects and their partners must agree to use a highly effective method of contraception. Effective birth control includes hormonal contraception (oral, intravaginal, transdermal, injectable or implantable), intrauterine device (IUD) plus one barrier method; or 2 barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm). Vasectomy (at least 3 months before IMP administration) and vasectomized partner (provided that the partner is the sole sexual partner of the trial participant and that the absence of sperm in the ejaculate has been confirmed) are acceptable methods of contraception, as well as post-menopausal female for at least 1 year (confirmed with serum follicle stimulating hormone [FSH] > 25.8 IU/L at screening), or surgically sterilized female subjects. Abstinence is not an acceptable contraception method. Female subjects who are of non-childbearing potential due to a surgical procedure or medical condition must provide documentation, and vasectomized male subjects must bring in the surgical report of the procedure.
6. Able to sign and understand an ICF and able to comply with study restrictions prior to selection.

Exclusion Criteria:

1. Presence or history of any disorder that may prevent the successful completion of the study.
2. Clinically significant abnormalities in laboratory test results (including hepatic and renal panels, complete blood count, chemistry panel and urinalysis), such as:

   * White blood cell count < 3.0x109/L.
   * Neutrophils < 1.5x109/L or clinically abnormal according to the subject's ethnic group (must be > 1.0x109/L for subjects of African descent).
   * Hemoglobin < 10 g/dL.
   * Platelet count < 125x109/L or > 450x109/L.
   * ALT > 1.5 ULN.
   * AST > 1.5 ULN.
   * Total bilirubin > 1.5 ULN (except in the presence of Gilbert's syndrome).
   * Creatinine > 1.2 ULN.
   * Sodium < 132 mmol/L or > 147 mmol/L.
   * Potassium < 3.2 mmol/L or > 5.5 mmol/L.
   * Chloride < 93 mmol/L or > 111 mmol/L.
   * Calcium < 8.3 mmol/L or > 10.7 mmol/L. Clinically significant abnormal values for all other laboratory parameters are at the investigator's discretion.
3. Any surgical or medical condition that may interfere with the absorption, distribution, metabolism, or excretion of the investigational medicine product.
4. Any history of drug related hypersensitivity reaction.
5. Prior treatment with a monoclonal antibody.
6. Intercurrent illness as evidenced by, e.g., nausea, vomiting, fever, or diarrhea) within 7 days before D1.
7. History of drug abuse (habitual taking of addictive or illegal drugs) within 1 year before D1.
8. Consumption of any caffeine-containing products (e.g., coffee, tea, chocolate, or soda) or grapefruit-containing products or alcoholic beverages within 48 hours before D1 and until D7.
9. Any condition or disease detected during the medical interview / physical examination that would render the subject unsuitable for the study, place the subject at undue risk or interfere with the ability of the subject to complete the study in the opinion of the Investigator or his designee.
10. Frequent headaches and/or migraine, recurrent nausea and / or vomiting.
11. Female subjects who are pregnant, or breastfeeding.
12. Positive screen for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates, phencyclidine [PCP]) and breath alcohol test at screening or D-2.
13. Positive serology for hepatitis B or hepatitis C or human immunodeficiency viruses (HIV).
14. Positive SARS-CoV-2 RT-PCR.
15. Any condition detected at screening that may interfere with or bias the physical examinations to be performed during the study.
16. Any prescribed or over-the-counter medication or herbal products taken within 1 week prior to start of administration of IMP (D1) or within 6 times the elimination half-life of the medication prior to start of IMP intake (whichever is longer), except birth control as described in inclusion criterion number 5 in Section 6.1. Vitamin/mineral supplements and occasional use of acetaminophen is allowed up until 24 hours before dosing.
17. Participation in a clinical trial or use of an investigational drug within 30 days before randomization.
18. Any vaccination within 30 days before signature of informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Assessment of adverse events (AEs) and treatment emergent adverse events (TEAEs) | Through study completion, an average of 60 days
Injection site safety and tolerability assessment | Visit Day 1
  Site injection tolerability will be assessed by the Investigator using a 4-level score (none, mild, moderate, severe) after IV infusion and SC injection.
Clinical laboratory measurements - Hematology - hemoglobin | Visits Day 1 through Day 60
  Hemoglobin (g/dL)
Clinical laboratory measurements - Hematology - hematocrit | Visits Day 1 through Day 60
  Hematocrit (%)
Clinical laboratory measurements - Hematology - erythrocytes | Visits Day 1 through Day 60
  Erythrocytes
Clinical laboratory measurements - Hematology - white blood cell count | Visits Day 1 through Day 60
  White blood cell count with differential (neutrophils, basophils, eosinophils, lymphocytes, monocytes and platelets) (X10(3)/UL)
Clinical laboratory measurements - Blood chemistry - sodium | Visits Day 1 through Day 60
  Sodium (mmol/L)
Clinical laboratory measurements - Blood chemistry - potassium | Visits Day 1 through Day 60
  Potassium (mmol/L)
Clinical laboratory measurements - Blood chemistry - calcium | Visits Day 1 through Day 60
  Calcium (mg/dL)
Clinical laboratory measurements - Blood chemistry - chloride | Visits Day 1 through Day 60
  Chloride (mmol/L)
Clinical laboratory measurements - Blood chemistry - CO2 | Visits Day 1 through Day 60
  CO2 (mmol/L)
Clinical laboratory measurements - Blood chemistry - blood urea nitrogen | Visits Day 1 through Day 60
  Blood urea nitrogen (mg/dl)
Clinical laboratory measurements - Blood chemistry - creatinine | Visits Day 1 through Day 60
  creatinine (mg/dL), glucose, total proteins, triglycerides, total cholesterol, AST, ALT, gamma-glutamyltransferase, creatinine phosphokinase, albumin, alkaline phosphatase, and total bilirubin
Clinical laboratory measurements - Blood chemistry - glucose | Visits Day 1 through Day 60
  Glucose (mg/dL)
Clinical laboratory measurements - Blood chemistry - total proteins | Visits Day 1 through Day 60
  Total proteins (g/dL), triglycerides, total cholesterol, AST, ALT, gamma-glutamyltransferase, creatinine phosphokinase, albumin, alkaline phosphatase, and total bilirubin
Clinical laboratory measurements - Blood chemistry - triglycerides | Visits Day 1 through Day 60
  Triglycerides (mg/dL)
Clinical laboratory measurements - Blood chemistry - total cholesterol | Visits Day 1 through Day 60
  Total cholesterol (mg/dL)
Clinical laboratory measurements - Blood chemistry - AST | Visits Day 1 through Day 60
  AST (U/L)
Clinical laboratory measurements - Blood chemistry - ALT | Visits Day 1 through Day 60
  ALT (U/L)
Clinical laboratory measurements - Blood chemistry - Gamma-glutamyltransferase | Visits Day 1 through Day 60
  Gamma-glutamyltransferase (U/L)
Clinical laboratory measurements - Blood chemistry - Creatinine phosphokinase | Visits Day 1 through Day 60
  Creatinine phosphokinase (mg/dL)
Clinical laboratory measurements - Blood chemistry - albumin | Visits Day 1 through Day 60
  Albumin (g/dL)
Clinical laboratory measurements - Blood chemistry - alkaline phosphatase | Visits Day 1 through Day 60
  Alkaline phosphatase (U/L)
Clinical laboratory measurements - Blood chemistry - total bilirubin | Visits Day 1 through Day 60
  Total bilirubin (mg/dl)
Clinical laboratory measurements - Coagulation - partial thromboplastin time | Visits Day 1 through Day 60
  Activated partial thromboplastin time (secs)
Clinical laboratory measurements - Coagulation - prothrombin time | Visits Day 1 through Day 60
  Prothrombin time (sec)
Clinical laboratory measurements - Coagulation - International normalized ratio | Visits Day 1 through Day 60
  International normalized ratio
Clinical laboratory measurements - Hormonology | Visits Day 1 through Day 90
  Measured parameters: Hormonology (TSH, FSH (for post-menopausal women); β-HCG (for women of childbearing potential))
Clinical laboratory measurements - Hormonology - TSH | Visits Day 1 through Day 90
  TSH (mIU/mL)
Clinical laboratory measurements - Hormonology - FSH | Visits Day 1 through Day 90
  FSH (mIU/mL)
Clinical laboratory measurements - Urinalysis - pH | Visits Day 1 through Day 60
  pH
Clinical laboratory measurements - Urinalysis - protein | Visits Day 1 through Day 60
  Protein (negative/positive)
Clinical laboratory measurements - Urinalysis - glucose | Visits Day 1 through Day 60
  Glucose (negative/positive)
Clinical laboratory measurements - Urinalysis - leukocytes | Visits Day 1 through Day 60
  Leukocytes (negative/positive)
Clinical laboratory measurements - Urinalysis - nitrites | Visits Day 1 through Day 60
  Nitrites (negative/positive)
Clinical laboratory measurements - Urinalysis - ketones | Visits Day 1 through Day 60
  Ketones (negative/positive)
Clinical laboratory measurements - Urinalysis - blood | Visits Day 1 through Day 60
  Blood (negative/positive)
Vital signs measurements - Blood pressure | Visits Day 1 through Day 90
  Supine and standing systolic and diastolic blood pressure (mmHg)
Vital signs measurements - Heart rate | Visits Day 1 through Day 90
  Heart rate (beats/min)
Vital signs measurements - Body temperature | Visits Day 1 through Day 90
  Body temperature (degrees Celsius)
Vital signs measurements - Respiratory rate | Visits Day 1 through Day 90
  Respiratory rate (breaths/min)
Electrocardiogram (ECG) measurements - Mean heart rate | Visits Day 1 through Day 90
  ECG mean heart rate (beats/min)
Electrocardiogram (ECG) measurements - PR interval | Visits Day 1 through Day 90
  PR interval, aggregate (msec)
Electrocardiogram (ECG) measurements - QRS axis | Visits Day 1 through Day 90
  QRS axis (deg)
Electrocardiogram (ECG) measurements - QTcF interval | Visits Day 1 through Day 90
  QTcF interval, aggregate (msec)

SECONDARY OUTCOMES:
Serum PK of single dose AV-380 via intravenous infusion and subcutaneous injection | Visits Day 1 through D90
  Cmax (maximum observed serum concentration)
Serum PK of single dose AV-380 via intravenous infusion and subcutaneous injection | Visits Day 1 through Day 90
  Tmax (time to reach maximum serum concentration)
To correlate the serum level of GDF-15 with the dose and serum level of AV-380 | Visits Day 1 through Day 90
  Emax (maximum effect observed)
To correlate the serum level of GDF-15 with the dose and serum level of AV-380 | Visits Day 1 through Day 90
  AUEC (area under the effect-time curve)
To correlate the serum level of GDF-15 with the dose and serum level of AV-380 | Visits Day 1 through Day 90
  TEmax (time to reach maximum effect)
AV-380 immunogenicity in healthy subjects - anti-AV-380 antibodies (human anti-human antibodies [HAHA]) levels in serum. | Visits Day 1 through Day 180
  HAHA levels
AV-380 immunogenicity in healthy subjects - Monocyte chemoattractant protein 1 (MCP-1) levels in serum. | Visits Day 1 and Day 2
  Serum MCP-1 levels will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Biotrial Inc., Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No